CLINICAL TRIAL: NCT00048672
Title: Therapy of Early Chronic Phase Chronic Myelogenous Leukemia (CML) With Gleevec (STI571)
Brief Title: Therapy of Early Chronic Phase CML With Gleevec
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-015
Record Dates: First submitted 2002-11-05; First posted 2002-11-06 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Leukemia, Myeloid, Chronic-Phase
Keywords: Early Chronic Phase Chronic Myelogenous Leukemia; Leukemia; Gleevec; STI571; Imatinib mesylate
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gleevec (Experimental): Gleevec 400 mg orally daily. Dose adjustments made at discretion of treating physician within these guidelines: The highest dose acceptable is 800 mg daily. The lowest dose acceptable is 300 mg. No dose adjustment of more than 200 mg at one time is allowed. Dose adjustments to less than 300 mg may be approved after consultation with the principal investigator.
  Interventions: Drug: Gleevec

INTERVENTIONS:
Drug: Gleevec — Starting dose of 400 mg orally daily.
  Other Names: Imatinib Mesylate; STI-571

SUMMARY:
The goal of this clinical research study is to see if imatinib mesylate (Gleevec, STI571) can improve CML in chronic phase.

Objectives:

Primary Objective:

To increase the proportion of patients achieving a complete cytogenetic response in patients with Ph-positive early chronic phase CML using initial Gleevec therapy.

Secondary Objective:

To evaluate the duration of cytogenetic response, duration of hematologic response and survival.

DETAILED DESCRIPTION:
Before treatment starts, patients will have a physical exam including medical history and documentation of disease, blood tests, and a bone marrow study. The bone marrow will be removed with a large needle.

Patients on this study will take 400 mg of imatinib daily (morning or evening). If you have side effects, the dose may be lowered. If the response is not good, the dose of imatinib mesylate will be increased to 800 mg daily (400 mg in the morning and 400 mg in the evening) or may be decreased to 300 mg daily based on how the drug is tolerated. Imatinib mesylate should be taken with a large glass of water. Bottles containing the tablets will be given to the patient every 6 months. Unused supplies must be returned at the end of the study.

After completing 3 to 12 months of therapy, response to imatinib mesylate will be evaluated. If the response is good, treatment with imatinib mesylate alone will be continued. Treatment may be continued for up to 20 years, or as long as it is judged best to control the leukemia.

Update: June 2010:

Blood tests are recommended 2 times per year. Your doctor will discuss with you how often you should have blood tests. Bone marrow will be done if your doctor thinks it is necessary to check your disease. You must return to MD Anderson at least once every year. You may not need a bone marrow test every visit, but you will have blood drawn to measure the amount of disease you have. If the leukemia cannot be found for 2 years or longer on the blood test called PCR which is done to measure the amount of disease you have, your doctor may talk to you about stopping treatment with imatinib. If you and your doctor decide to stop your therapy, you will have a blood test for PCR done every 3 to 6 months. You do not need to return to MD Anderson to have this blood test done. You may have the blood taken by your local doctor and mailed to MD Anderson. If the leukemia is found again by the PCR blood test, your doctor may recommend that you restart treatment with imatinib. You may decide to stay on treatment with imatinib even if your PCR blood test does not show any sign of leukemia for 2 years or longer.

This is an investigational study. Imatinib mesylate has been approved in CML. A total of 50 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Philadelphia chromosome (Ph)- positive or breakpoint cluster region (bcr)-positive CML in early chronic (diagnosis < 12 months).
2. Age 15 years or above
3. Adequate renal, hepatic, cardiac and performance status (ECOG 0-2) - no psychiatric disability (psychosis)
4. Signed informed consent

Exclusion Criteria:

1. Grade 3-4 cardiac
2. Psychiatric problem
3. Pregnant or lactating

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2001-03; Primary Completion 2002-11 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of patients achieving complete cytogenetic response using initial Gleevec therapy | Baseline to 12 Months

SECONDARY OUTCOMES:
Duration of cytogenic response, hematologic response and survival | Baseline, 12 Months, 2 Years or until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jain P, Kantarjian H, Boddu PC, Nogueras-Gonzalez GM, Verstovsek S, Garcia-Manero G, Borthakur G, Sasaki K, Kadia TM, Sam P, Ahaneku H, O'Brien S, Estrov Z, Ravandi F, Jabbour E, Cortes JE. Analysis of cardiovascular and arteriothrombotic adverse events in chronic-phase CML patients after frontline TKIs. Blood Adv. 2019 Mar 26;3(6):851-861. doi: 10.1182/bloodadvances.2018025874. PMID 30885996
- [Derived] Issa GC, Kantarjian HM, Gonzalez GN, Borthakur G, Tang G, Wierda W, Sasaki K, Short NJ, Ravandi F, Kadia T, Patel K, Luthra R, Ferrajoli A, Garcia-Manero G, Rios MB, Dellasala S, Jabbour E, Cortes JE. Clonal chromosomal abnormalities appearing in Philadelphia chromosome-negative metaphases during CML treatment. Blood. 2017 Nov 9;130(19):2084-2091. doi: 10.1182/blood-2017-07-792143. Epub 2017 Aug 23. PMID 28835440
- [Derived] Jain P, Kantarjian H, Nazha A, O'Brien S, Jabbour E, Romo CG, Pierce S, Cardenas-Turanzas M, Verstovsek S, Borthakur G, Ravandi F, Quintas-Cardama A, Cortes J. Early responses predict better outcomes in patients with newly diagnosed chronic myeloid leukemia: results with four tyrosine kinase inhibitor modalities. Blood. 2013 Jun 13;121(24):4867-74. doi: 10.1182/blood-2013-03-490128. Epub 2013 Apr 25. PMID 23620574
- See also: M.D. Anderson's website — http://www.mdanderson.org